CLINICAL TRIAL: NCT05957939
Title: Targeting Triple-negative Breast Cancer or ER-positive, PR Positive her2 Negative by Alkaline Glucosodiene Molecules Via a Metabolic Pathway Phase I Clinical Trial
Brief Title: Targeting Metastatic Breast Cancers by Alkaline Glucosodiene Molecules Via a Metabolic Pathway Phase I Clinical Trial
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ministry of Health, Saudi Arabia (Other Government)
Collaborators: Maher M.akl (Unknown)
Responsible Party: Principal Investigator, Amr kamel khalil Ahmed, Director of tuberculosis mobile team, Ministry of Health, Saudi Arabia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Maher M.Akl, Amr Ahmed
Record Dates: First submitted 2023-06-19; First posted 2023-07-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: TNBC - Triple-Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: a case study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- a case study with TNBC or ER positive , PR positive HER2 negative , (Experimental): researchers will study a case with metastatic breast cancer stage 4 and the source of nutrition either glucose source as energy fuel of cells or another nutrition ( alkaline glucosodiene)
  Interventions: Drug: Alkaline Glucosodiene Molecules

INTERVENTIONS:
Drug: Alkaline Glucosodiene Molecules — Toxic chemotherapeutic nutrition of cancer cells by alkaline glucosodiene molecules via targeting metabolic of cancerous tumors: a promising treatment

SUMMARY:
The diverse group of breast tumors known as triple-negative breast cancer (TNBC) which is lethally and deadly type of breast cancer and insensitive to endocrine therapy and HER2-targeted therapy because it lacks the expression of estrogen, progesterone, and human epidermal growth factor receptors TNBC makes up almost 15% of all invasive breast cancers, and of all breast tumor subtypes, it has the worst overall survival and the highest rate of metastatic occurrence. Cytotoxic chemotherapy is the main established systemic therapy for early and advanced TNBC disease at the moment because there is no authorized targeted therapy. Despite the fact that chemotherapy greatly improves clinical outcomes for TNBC patients, recurrence rates are still high and TNBC cancers frequently develop chemotherapeutic drug resistance ). In light of the few available therapy choices, so few choices for this subtype of breast cancer, and many cases are resistant to chemotherapy and recurrent and with a risk of high metastasis from previous literature and many experimental studies, the target of glucose environment is a promising weapon against this deadly type of breast cancer so glucose deprivation from tumor cells may cut the glucose entry as fuel to these cancer cells so this study uses a substitute energy fuel by using alkaline glucosodiene which is chemically invented by Maher M.AKL

DETAILED DESCRIPTION:
Breast cancer is the most frequently diagnosed and the second largest cause of cancer-related deaths in women aged 29 to 59 worldwide[1-4]. It is a genetically heterogeneous illness. Breast cancer treatments available today may help increase patient survival. However, one-third of patients with aggressive triple-negative breast cancer (TNBC), which accounts for 17-20 percent of all breast cancers [5-7], may experience more relapses than patients with subtypes of breast cancer that express receptors for the hormones estrogen (ER), progesterone (PR), or human epidermal growth factor (HER-2). The 17-20 percent of TNBC patients who experience this eventually pass away from a distant metastatic disease[5, 8-10]. Although decades of research have improved our understanding of the issue, the pathobiology of breast cancer progression's basic mechanisms remain a mystery.Cancer is a genetic disease characterized by heritable defects in cellular regulatory mechanisms. Tumor cells must adapt their metabolism to survive and proliferate in the challenging conditions of the tumor microenvironment. To maintain uncontrolled cellular growth and survival, cancer cells alter their metabolism, which makes them dependent on a steady supply of nutrients and energy. Almost a century ago, the Warburg theory suggested that cancer cells consume glucose even in the presence of oxygen. Recent studies have confirmed that cancer cells indeed consume significantly more glucose than normal cells. Cancerous tumors require an acidic microenvironment with low oxygen levels for growth and spread. However, recent advances in pH measurement have shown that the intracellular pH of cancer cells is neutral or slightly alkaline compared to normal tissue cells. This finding indicates that not all tumors are highly acidic. Taking advantage of cancer cells' high glucose consumption, a strategy to lyse cancer cells is tested by means of glucose modifications that exploit the characteristics of their uncontrolled growth process.

From the study of the molecular structure to give him alkaline properties that enable him to make defects in the tumor structure and possibly achieve cell killing, this situation will have a killing effect on cancer cells if small molecules of toxic atoms (alkaline atoms) can be continuously supplied to them through food, due to the uncontrolled consumption of glucose molecules by cancer cells. This theory attempts to investigate by changing the atomic structure of glucose molecules to make them alkaline glucosodiene molecules as one of the methods to kill cancer cells. By preparing alkaline glucosodiene molecules and performing animal experiments and histological observations, it was shown that tumors without alkaline treatment showed a tendency to infiltrate and grow, while tumors treated with glucosodiene molecules showed complete disappearance of cell structure and nucleolysis, supporting the validity of the theory. Cancer cells are known to be more sensitive to heat and apoptosis than normal cells, and this property has been leveraged to develop glucosodiene molecules that induce tumor hyperthermia. The chemical mechanism of sodium processing in this approach is similar to the cathode reaction in electrochemotherapy. Cancer cells take up glucosodiene because they are capable of growing uncontrollably and lack the sophisticated brain function necessary to distinguish between glucose and modified glucose. Glucosodiene kills cancer cells by breaking down glucose molecules into carbon dioxide and water, generating energy that alkali elements utilize to dissolve cancer cells from within. This approach is effective for treating numerous types of cancer due to the uncontrolled development of cancer cells. The traditional approach of eliminating cancer cells is not applicable in this theory, as cancer cells are dissolved from within due to their uncontrollable consumption of glucose molecules. Cancer cells have an uncontrolled ability to multiply and consume glucose molecules. Glucosodiene molecules have been developed to exploit this characteristic by inducing tumor hyperthermia, which makes cancer cells more sensitive to heat and apoptosis. Glucosodiene breaks down glucose molecules into carbon dioxide and water, generating energy that is utilized by alkali elements to dissolve cancer cells from within. Cancer cells that consume sodium-laced glucose struggle to retain their rigid cell structure and instead disintegrate and dissolve into the bloodstream before being excreted as urine. This approach is particularly effective in treating numerous types of cancer because cancer cells predominantly grow in lumped form, allowing for a the localized concentration of alkali elements. so this clinical trial uses case with TNBC ( ) and studies the environment of the tumor at many different environments like high glucose, zinc, insulin, interleukin -6 .

Glucosodiene may hasten the death of aging cells, which resist elimination. The breakdown of sugar molecules without oxygen causes acid, but discomfort subsides when cells take up glucosodiene. The body's T cells eliminate any remaining cancer cells after recovery [28]. Normal cells can regulate their natural alkalinity and excrete excess pH [29, 30]. This could be a significant development in chemotherapy, with fewer side effects than conventional drugs. Further research is required. Ethical approval will apply to ethical committee at Mansoura university faculty of medicine

ELIGIBILITY:
Inclusion Criteria:

* Type of patient: Female patient
* Age: 18-55 years
* Type of breast cancer: metastatic breast cancer hormonal or triple-negative breast cancer

Exclusion Criteria:

* with other co-morbidities like diabetes or hypertension
* with other type of cancers
* on other chemotherapy or immunotherapy or hormonal therapy

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
the Progression-free survival (PFS) | Time Frame: 30 days after treatment
  the time from treatment initiation until disease progression or worsening may be used as a direct or surrogate measure of clinical benefit for drug approvals, depending on the disease and response observed
Disease-free survival (DFS) | Time Frame: 30 days after treatment
  time from treatment until the recurrence of disease (or death) after undergoing curative-intent treatment.

SECONDARY OUTCOMES:
the change in tumor size or fungating wound at the original site of tumor | Time Frame: 30 days after treatment
  researchers will register the changes either improvement or progression at the original wound after mastectomy and overall symptoms of metastatic patient like headache, body aches, vomiting , gaspings , salty taste

IPD SHARING:
Plan to Share IPD: Yes